CLINICAL TRIAL: NCT05761314
Title: Incidence and Molecular Pathogenesis of Solid Tumors in RASopathies
Brief Title: Solid Tumors in RASopathies
Acronym: 4218
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4218
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: RASopathy; Costello Syndrome; Cardio-Facio-Cutaneous Syndrome; Noonan Syndrome
MeSH Terms: conditions — Costello Syndrome; Cardiofaciocutaneous syndrome; Noonan Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Case group (Experimental): To report the prevalence of solid tumors in a monocentric cohort of individuals with RASopathies
  Interventions: Diagnostic Test: Molecular characterization of solid tumor in RASopathies

INTERVENTIONS:
Diagnostic Test: Molecular characterization of solid tumor in RASopathies — NGS analysis on tumor sample

SUMMARY:
RASopathies are a group of syndromes, caused by variants of genes involved in the regulation of the Ras/MAP/ERK pathway. This intracellular transduction pathway profoundly affects embryogenic development, organogenesis, synaptic plasticity and neuronal growth.

RASopathies are characterized by multi-organ involvement, growth delay, premature aging and haemato-oncological manifestations.

Based on evidences provided by literature, cancer screening protocols are applied in some individuals affected by RASopathies, even though detailed information about prevalence and molecular pathogenesis of such tumors is still not clearly elucidate.

DETAILED DESCRIPTION:
To define the prevalence of solid (non-haematological) neoplasms in a monocentric cohort of patients affected by RASopathies To perform Next Generation Sequencing (NGS) analysis on tissue samples to preliminarily characterize the molecular pathogenesis of solid tumors in these patients' categories.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and molecularly confirmed diagnosis of a RASopathy

Exclusion Criteria:

* Clinical diagnosis of RASopathy without molecular characterization

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2026-10-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of solid tumors in RASopathies | 5 years
  To detect prevalence of solid tumors in monocentric cohort of RASopathies

SECONDARY OUTCOMES:
Molecular characterization of solid tumors in RASopathies | 5 years
  NGS analysis on tumor tissue samples

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Leoni, MD, PhD, Principal Investigator — Fondazione Policlinico A. Gemelli, IRCCS
Locations (1):
- Department of Woman and Child Health and Public Health, Fondazione Policlinico A. Gemelli, IRCCS, Roma, Italy